CLINICAL TRIAL: NCT04170569
Title: The Effect of Yoga on Posttraumatic Growth and Quality of Life in the Postpartum Period
Brief Title: Yoga on Posttraumatic Growth and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Hacer Unver, PhD, Inonu University, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Inonu University.
Record Dates: First submitted 2019-10-29; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Posttraumatic Growth; Quality of Life
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Randomized Controlled trial with a prospective pretest-posttest experimental model
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Yoga program was applied.
  Interventions: Behavioral: Yoga
- Control Group (No Intervention): No yoga program.

INTERVENTIONS:
Behavioral: Yoga — Yoga Practice and Program: Yoga practice consisted of 10 weeks. Yoga practice involved following stages; 5-minute breathing exercises in standing or sitting position, 40-minute postpartum period specific asanas and last 15- minute deep relaxation in lying position were made by the researcher.
  Arms: Experimental Group

SUMMARY:
The objective of this study is to examine the effect of yoga on posttraumatic growth and quality of life. The birth action, which includes positive and negative experiences, can be an important opportunity to achieve posttraumatic growth and improve the quality of life.

This is a experimental model with pretest-posttest control group study. Two hundred and fifty-two women who met the criteria for inclusion in the study made up the research population. Three instruments were used to obtain the research data: Personal Information Form, Posttraumatic Growth Inventory (PTGI) and SF-36 Quality of Life Questionnaire (SF-36).

DETAILED DESCRIPTION:
Failure in modern medicine approaches or side effects of treatments and drugs, as well as the woman's anxiety to hurt herself and her baby direct her and her relatives to try complementary therapies. Women should prefer natural ways in coping with these postpartum problems rather than seeking medical advice.

When yoga and meditation, which are included in the group of mind-body-based complementary therapies, are performed in the postpartum period, they will help to relieve tensions and distresses that accumulate during birth, strengthen the pelvic floor, heal perineum, bring reproductive organs back to their prepregnancy condition healthily, provide the mother and the infant a sleep pattern, and have an easier transition to sleep.

ELIGIBILITY:
Inclusion Criteria:

* Having a baby between 2 and 6 months
* First time mom
* No tissue deformity in extremities

Exclusion Criteria:

* Any gynecological disease
* Any psychiatric illness
* Using any psychiatric medication

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — it is a study specific to postpartum period.
Enrollment: 80 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2019-01-19 (Actual)

PRIMARY OUTCOMES:
The Effect of Yoga on Posttraumatic Growth in the Postpartum Period | 10 weeks
  The posttraumatic growth scale for measure posttraumatic growth;The scale is scored from 0 to 5 and the lowest is 0 and the highest is 105. The higher the scores obtained, the higher the approval from the traumatic experience shows that it is experiencing high growth. There are three sub-dimensions: the change in self-perception of the scale, the change in philosophy of life, and the change in relationship with others.
The Effect of Yoga on Quality of Life in the Postpartum Period | 10 weeks
  SF-36 Quality of life scale for measure the quality of life; The scale is calculated by inverting the items 1, 6, 7, 8, 9d, 9e, 9h, 11b, 11d. Total score is not calculated in the scale. The subscales evaluate health between 0-100 points. 0 indicates "poor health" and 100 indicates "good health.Higher scores obtained from the subscales of the scale indicate that the quality of life level is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacer, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No